CLINICAL TRIAL: NCT03036878
Title: Evaluation of the ReNu™ Amniotic Suspension Allograft After Marrow Stimulation in the Treatment of Osteochondral Defects
Brief Title: ReNu™ Marrow Stimulation Augmentation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed for lack of enrollment
Sponsor: NuTech Medical, Inc (Industry)
Collaborators: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD-2016-04-02
Record Dates: First submitted 2017-01-27; First posted 2017-01-30 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Osteochondral Defect
Keywords: Osteochondral; Marrow Stimulation; ReNu

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ReNu Injection (Experimental): Injection of ReNu allograft into the joint capsule.
  Interventions: Other: ReNu

INTERVENTIONS:
Other: ReNu — ReNu is an allograft tissue composed of particularized amniotic membrane and cell from the amniotic fluid.

SUMMARY:
To evaluate the use of ReNu™ allograft for the augmentation of marrow stimulation for osteochondral lesions

DETAILED DESCRIPTION:
This is a prospective, non-randomized, longitudinal study of up to 8 evaluable participants recruited from two separate practices. Male and non-pregnant female patients between the ages of 18 and 55 years of age will be screened for study recruitment. Female patients must be actively practicing a contraception method, abstinence, be surgically sterilized, or be postmenopausal. Participants will receive ReNu™ as an adjunct to their standard of care marrow stimulation for the treatment of osteochondral defects.

At each follow-up visit, concomitant medications and adverse events shall be collected from each subject, and each subject shall complete the following questionnaires:

IKDC Health Assessment (Includes Short Form-36) Tegner KOOS Knee Survey VAS Pain Scale SANE score

The subjects will be assessed at Baseline using these scales an again at all subsequent study follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signature of the IRB approved Informed Consent
2. Male or female participants between the ages of 18-55
3. If female:

   1. Actively practicing a contraception method, or
   2. Practicing abstinence, or
   3. Surgically sterilized, or
   4. Postmenopausal
4. Pretreatment arthroscopic confirmation indicating one or two contained lesion(s) and equal to an ICRS Grade 3a, 3b, 3c, 3d of the femoral condyle, patella, or trochlear groove and OCD lesions (Grade 4a) with healed bone base, which is non-sclerotic and no loss of bone greater then 6mm measured from the surrounding subchondral plate. Original pretreatment arthroscopic confirmation indicates that one or two lesion(s) are equal to an ICRS Grade 3a, 3b, 3c, 3d contained lesion(s) that is equivalent to an Outerbridge Grade III or IV (greater than 50% loss of articular cartilage). OF NOTE: Patients with need for concomitant procedures such as Anteromedialization of Tibial Tubercle (AMZ) and lateral lengthening are allowable
5. Has peripheral cartilage debridement to healthy cartilage that results in a lesion (s) with an area of > or = 1cm ^2 and < or = 4 cm^2.
6. PCL, LCL and MCL in the affected knee are stable and the ACL is stable or can be stabilized as a concomitant procedure.
7. Ipsilateral knee compartment has intact menisci (or requires partial meniscectomy resulting in stable menisci). Minimum remnant width of 5mm.
8. The contralateral knee is asymptomatic, stable, and fully functional.
9. Must be physically and mentally willing and able to comply with post-operative rehabilitation and routinely scheduled clinical and radiographic visits through 24 months.
10. Alignment: Mechanical axis must be no more than 5 degrees from neutral.
11. Must be 3 months post previous surgery.

Exclusion Criteria:

1. Clinical and/or radiographic disease diagnosis of the indexed affected joint that Includes:

   1. Osteoarthritis or avascular necrosis,
   2. Rheumatoid arthritis, or history of septic or reactive arthritis,
   3. Gout or history of gout or pseudogout in the affected knee,
   4. Osteochondritis dissecans of the knee with significant bone loss (greater than 6mm deep from the subchondral plate)
   5. Associated damage to the underlying subchondral bone requiring a bone graft
2. History of secondary arthropathies (i.e. sickle cell disease, hemochromatosis, or autoimmune disease).
3. Uncontrolled diabetes.
4. Displays a high surgical risk due to unstable cardiac and/or pulmonary disease.
5. Has HIV or other immunodeficient state including subjects on immunosuppressant therapies, or has significant illness (metastasis of any type) that decreases the probability of survival to the 2 year endpoint.
6. Is at substantial risk for the need of organ transplantation, such as renal insufficiency.
7. Is pregnant or breast-feeding.
8. Body mass index > 35.
9. Has bipolar articular cartilage involvement or kissing lesions of the ipsilateral compartment, described as tibial or patellar lesions in the same compartment with greater than ICRS Grade 2 chondrosis.
10. Is participating concurrently in another clinical trial, or has participated in a clinical trial within 30 days of surgery.
11. Is receiving prescription pain medication other than NSAIDs or acetaminophen for conditions unrelated to the index knee condition, chronic use of anticoagulants, or taking corticosteroids.
12. Has a neuromuscular, neurosensory, or musculoskeletal deficiency that limits the ability to perform objective functional assessment of either knee.
13. Active joint infection.
14. Prior total meniscectomy of either knee.
15. Radiographically has >5 degrees of malalignment as measured from the hip, knee and ankle mechanical axis.
16. Has subchondral bone loss of greater than 6mm
17. Has received within the past three months intra-articular platelet rich plasma, hyaluronic acid therapy, steroid, amniotic-derived or stem cell injections in the index knee.
18. Prior realignment surgery in the affected knee within the past 6 months.
19. Failed microfracture/marrow stimulation treatment performed less than 12-months before baseline.
20. Is receiving workman's compensation or currently involved in litigation relating to the index knee.
21. Has history of alcoholism, medication, or intravenous drug abuse, psychosis, is a prisoner, has a personality disorder (s), poor motivation, emotional or intellectual issues that would likely make the subject unreliable for the study, or any combination of variables in the investigator's judgment that should exclude a potential subject.
22. Any conditions or implants that might affect having MRIs: had or have an aneurysm clip implanted, intraocular foreign bodies (commonly seen in welders), subcutaneous metal shards (found in sheet metal workers), or some shrapnel; additionally, no cardiac pacemaker, defibrillator, implanted neurostimulater (TENS implants) some prosthetic heart valve (especially mitral valve), cochlear implant or other hearing aide. Subjects should be excluded if they have a tendency of claustrophobia or have tattoos that may contain iron-based dyes.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Change in KOOS score from baseline | 1 Year
Change in Tegner score from baseline | 1 Year

SECONDARY OUTCOMES:
Change in VAS score from baseline | 6, 12 & 24 months
Change in Tegner score from baseline | 6 & 24 months
Change in SANE score from baseline | 6, 12 & 24 months
Change in KOOS score from baseline | 6 & 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jack Farr, MD, Principal Investigator — OrthoIndy
Locations (2):
- United States (2):
  - Orthoindy, Indianapolis, Indiana
  - Hospital for Special Surgery, New York, New York

IPD SHARING:
Plan to Share IPD: No